CLINICAL TRIAL: NCT02845804
Title: Harmonizing Optimal Strategy for Treatment of Coronary Atherosclerotic Lesions- Registry-based Study on the Effect and Safety of Xience Xpedition™/Alpine™, Everolimus-eluting Stent for Coronary Atherosclerotic Lesions: HOST-Alpine Registry
Brief Title: Effect and Efficacy of Xpedition™/Alpine™, Everolimus-eluting Stent for Coronary Atherosclerosis
Acronym: HOST-ALPINE
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Seoul National University Hospital (Other)
Collaborators: Abbott (Industry)
Responsible Party: Principal Investigator, Hyo-Soo Kim, Professor, Seoul National University Hospital
Other Study IDs: HOST-ALPINE
Record Dates: First submitted 2016-07-24; First posted 2016-07-27 (Estimated); Last update posted 2016-07-27 (Estimated); Status verified 2016-07

CONDITIONS: Coronary Artery Disease; Percutaneous Coronary Intervention; Acute Coronary Syndrome; Angina Pectoris
Keywords: coronary artery disease; percutaneous coronary intervention; everolimus-eluting stents
MeSH Terms: conditions — Coronary Artery Disease; Acute Coronary Syndrome; Angina Pectoris

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Alpine: The patients who received percutaneous coronary intervention with Xience Xpedition™/Alpine™
  Interventions: Device: Alpine

INTERVENTIONS:
Device: Alpine
  Other Names: Everolimus-eluting stent

SUMMARY:
The objectives of this study are

1. To establish a prospective registry of the whole patients who received percutaneous coronary intervention with Xience Xpedition™/Alpine™ stent
2. To evaulate the long-term efficacy and safety of coronary stenting with the Xience Xpedition™/Alpine™ stent
3. To compare the long-term efficacy and safety of coronary stenting between the Xience Xpedition™/Alpine ™ stent and other contemporary drug-eluting stents which had established their own registry

DETAILED DESCRIPTION:
Secondary endpoints of this study are

Stent thrombosis-24 hours(acute), 30 days(subacute), 1 year(late), every 1 year till 3 years(very-late) after index PCI

Target vessl failure

Composite rate of cardiac death and any MI, 3 years

Composite rate of all death and any MI

Composite rate of all death, any MI, and any repeat revascularization

Compliance and therapy interruptions with prescribed adjunctive antiplatelet therapy

ELIGIBILITY:
Inclusion Criteria:

* The patient agrees to participate in this study by signing the informed consent form.

Alternatively, a legally authorized patient representative may agree to the patient's participation in this study and sign the informed consent form

Exclusion Criteria:

* There are no exclusion criteria for this registry.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All coronary arterial disease patients who received percutaneous coronary intervention with Xience Xpedition™/Alpine™ stent(s)
Sampling Method: Non-Probability Sample
Enrollment: 1533 (Estimated)
Dates: Start 2015-07; Primary Completion 2018-07 (Estimated); Study Completion 2021-07 (Estimated)

PRIMARY OUTCOMES:
Target lesion failure | 12 months
  Composite of cardiac death, non-fatal target vessel-related myocardial infarction (MI), and ischemia-driven target lesion revascularization (TLR)

SECONDARY OUTCOMES:
Target vessel failure | 12 months
  Composite of cardiac death, non-fatal target vessel related myocardial infarction, and ischemia-driven target vessel revascularization (TVR)
Composite rate of cardiac death and myocardial infarction | 12 months, 3 years
Composite rate of all-cause death and any myocardial infarction | 12 months, 3 years
Composite rate of all-cause death and any myocardial infarction, and any repeat revascularization | 12 months, 3 years
Rate of compliance and interruptions with prescribed adjunctive antiplatelet therapy | 12 months, 3 years
Clinical device and procedural success rate | intraoperative
Stent thrombosis | within 24 hours, 1 - 30 days, 31 days - 1 year, after 1 year
  acute (within 24 hours), subacute (1 - 30 days), late (31 days - 1 year), very late (>1 year)

CONTACTS AND LOCATIONS:
Overall Officials: Hyo-soo Kim, MD, PhD, Study Chair — Seoul National University Hospital
Locations (20):
- South Korea (20):
  - Kangwon National University Hospital, Chuncheon, Gangwon-do
  - Wonju Severance Christian Hospital, Wŏnju, Gangwon-do
  - Sejong General Hospital, Bucheon-si, Gyeonggi-do
  - Hallym University Sacred Heart Hospital, Anyang
  - Busan Paik Hospital, Busan
  - Kosin University Gospel Hospital, Busan
  - Dankook University Hospital, Cheonan
  - SoonChunHyang University Cheonan Hospital, Cheonan
  - Yongnam University Medical Center, Daegu
  - Chonnam National University Hospital, Gwangju
  - Wonkwang University Hospital, Iksan
  - Inha University Hospital, Inchon
  - Chungbuk National University Hospital, Jeonju
  - Presbyterian Medical Center, Jeonju
  - Seoul National University Bundang Hospital, Seongnam
  - Gangbuk Samsung Hospital, Seoul
  - Hanyang University Medical Center, Seoul
  - Kangdong Sacred Heart Hospital, Seoul
  - Seoul Boramae Hospital, Seoul
  - Seoul National University Hospital, Seoul